CLINICAL TRIAL: NCT00669084
Title: Studies of Innate and Acquired Resistance to P. Falciparum Malaria in Mali
Brief Title: Innate and Acquired Resistance to Plasmodium Falciparum Malaria in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908120; 08-I-N120
Record Dates: First submitted 2008-04-26; First posted 2008-04-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-11-19

CONDITIONS: Malaria
Keywords: Innate Immunity; Malaria; Plasmodium; Hemoglobinopathy; G6PD Deficiency
MeSH Terms: conditions — Malaria; Hemoglobinopathies; Glucosephosphate Dehydrogenase Deficiency

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, sponsored by NIAID and the University of Bamako, Mali, will identify genetic and other factors that may protect against severe malaria in some children.

Children between 6 months and 17 years of age who live in Kenieroba, Fourda or Bozokin villages in Mali may enroll in the study. Participants have a blood sample collected by finger prick with a small needle. The blood is examined for gene variants that influence the severity of disease in children exposed to the malaria parasite.

Children who develop a fever or other symptoms of malaria are evaluated and treated in Kenieroba s health center for up to 5 years from entering the study, or until they reach 18 years of age. The children are treated with artesunate and amodiaquine. Children with severe disease are treated with quinine. One tablespoon of blood is drawn from the children for study.

At the end of the dry season and the wet season, a subset of 200 healthy children are asked to provide 1 or 2 tablespoons of blood, drawn through a needle placed in a vein in the arm. Additional research blood samples may be requested from children between 2 and 17 years old. Blood will not be taken from any child more than twice a year.

...

DETAILED DESCRIPTION:
Hemoglobin (Hb) and red blood cell (RBC) polymorphisms that give rise to HbS, HbC, alpha-thalassemia, G6PD-deficiency, and ABO blood groups occur at high frequency in Mali. To determine whether these Hb/RBC polymorphisms are associated with protection against mild malaria and malaria-associated anemia, we will conduct a cohort study in Mali. Approximately 1300 children will be genotyped for five Hb/RBC polymorphisms and followed for 5 years to compare mean incidence rates for mild malaria, stratified by polymorphism. Differences between Hb levels during acute malaria episodes and at baseline will be calculated to determine if Hb/RBC polymorphisms influence the degree of malaria-associated anemia. To investigate whether Hb/RBC polymorphisms impair monocyte activation, we will obtain parasites from children with malaria, culture them in RBCs of different genotype, and compare the parasitized RBCs for their ability to activate monocytes in vitro. Plasma samples from children with malaria will also be compared for their levels of monocyte-derived cytokines. A variety of single nucleotide polymorphisms (SNPs) in immune response genes have recently been identified in African populations. To determine whether these polymorphisms are associated with protection against severe malaria, we will compare the prevalence of SNPs in groups of children with severe or mild malaria. Blood Collection Study. Components of the innate immune system (e.g., Toll-like receptors) expressed on antigen presenting cells (APC) provide the first line of defense against microbial infection and frame the nature and scale of adaptive immune responses. To investigate whether APC from malaria-experienced individuals respond to TLR ligands in vitro stimulation assays, we will obtain blood samples from 100 healthy children in the dry season and again in the wet season. Immunological memory is a key feature of adaptive immunity and involves memory T cells. Clinical trials in which malaria-nafve human volunteers were vaccinated with merozoite MSP-1 antigens enabled us to study the development of immunological memory by measuring memory T cell cytokine production and expression of surface activation markers. To investigate whether memory T cells from malaria-experienced individuals respond similarly to AMA-I/MSP-1 ligands in vitro stimulation assays, we will obtain blood samples from an additional 100 healthy children in the dry season and again in the wet season. These collections of paired samples will enable us to explore the possibility that TLR- and AMA-1/MSP-l-induced immune responses are boosted during a transmission season and increase with age (a surrogate for disease controlling immunity).

ELIGIBILITY:
* INCLUSION CRITERIA:

(Cohort Study)

* Resident of Kenieroba, Fourda, or Bozokin villages, and no plans to relocate away from the study village for the next 5 years.
* Willingness to participate in the study as evidenced by informed consent of parents or guardians of children, and willingness to bring children to study clinic if they develop fever or other symptoms of malaria.
* Age 6 months to 17 years.

(Blood Collection Study)

* Children enrolled in the cohort study.
* Willingness to participate in the study as evidenced by informed consent of parents or guardians of children.
* Age 2 years to 14 years.
* Hemoglobin level greater than or equal to 8.5g/dL.

(Parasite Clearance Study)

* Children enrolled in the cohort study.
* Willingness to participate in the study as evidenced by informed consent of parents or guardians of children.
* Age 1 year to 17 years (inclusive).
* P. falciparum density greater than or equal to 10,000/microL.
* Present with their first episode of uncomplicated malaria of the 2010 transmission season or any episode during the 2012 transmission season.
* Resident of Kenieroba

(Adult blood Collection Study)

* Willingness to participate in the study as evidenced by informed consent.
* Age 18 years to 65 years.
* Hemoglobin level greater than or equal to 8.5 g/dL

EXCLUSION CRITERIA:

(Cohort Study)

* Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric disease).
* Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS) or to the child (e.g., severe malnutrition).

(Blood Collection Study)

* Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric disease).
* Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS) or to the child (e.g., severe malnutrition).

(Parasite Clearance Study)

* Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric diesase).
* Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS) or to the child (e.g., severe malnutrition).
* Pregnancy at the time of malaria episode.

(Adult Blood Collection Study)

* Any condition that in the opinion of the investigator would render the subject unable to comply with the protocol (e.g., psychiatric disease)
* Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary exposure risks to study personnel (e.g., individuals who are known to be HIV-infected or to have AIDS.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1718 (Actual)
Dates: Start 2008-04-21; Study Completion 2013-11-19

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Odontostomatology, Bamako, Mali

REFERENCES:
- [Background] Fairhurst RM, Baruch DI, Brittain NJ, Ostera GR, Wallach JS, Hoang HL, Hayton K, Guindo A, Makobongo MO, Schwartz OM, Tounkara A, Doumbo OK, Diallo DA, Fujioka H, Ho M, Wellems TE. Abnormal display of PfEMP-1 on erythrocytes carrying haemoglobin C may protect against malaria. Nature. 2005 Jun 23;435(7045):1117-21. doi: 10.1038/nature03631. PMID 15973412
- [Background] Guindo A, Fairhurst RM, Doumbo OK, Wellems TE, Diallo DA. X-linked G6PD deficiency protects hemizygous males but not heterozygous females against severe malaria. PLoS Med. 2007 Mar;4(3):e66. doi: 10.1371/journal.pmed.0040066. PMID 17355169
- [Background] Luzzatto L, Usanga FA, Reddy S. Glucose-6-phosphate dehydrogenase deficient red cells: resistance to infection by malarial parasites. Science. 1969 May 16;164(3881):839-42. doi: 10.1126/science.164.3881.839. PMID 4889647
- [Derived] Suresh RV, Deng B, Gebremicale Y, Roche K, Miura K, Long C. Mesenchymal stem cells of the bone marrow raise infectivity of Plasmodium falciparum gametocytes. mBio. 2023 Dec 19;14(6):e0223223. doi: 10.1128/mbio.02232-23. Epub 2023 Nov 1. PMID 37909740
- [Derived] Lopera-Mesa TM, Doumbia S, Konate D, Anderson JM, Doumbouya M, Keita AS, Diakite SA, Traore K, Krause MA, Diouf A, Moretz SE, Tullo GS, Miura K, Gu W, Fay MP, Taylor SM, Long CA, Diakite M, Fairhurst RM. Effect of red blood cell variants on childhood malaria in Mali: a prospective cohort study. Lancet Haematol. 2015 Apr;2(4):e140-9. doi: 10.1016/S2352-3026(15)00043-5. Epub 2015 Mar 24. PMID 26687956
- [Derived] Lopera-Mesa TM, Doumbia S, Chiang S, Zeituni AE, Konate DS, Doumbouya M, Keita AS, Stepniewska K, Traore K, Diakite SA, Ndiaye D, Sa JM, Anderson JM, Fay MP, Long CA, Diakite M, Fairhurst RM. Plasmodium falciparum clearance rates in response to artesunate in Malian children with malaria: effect of acquired immunity. J Infect Dis. 2013 Jun 1;207(11):1655-63. doi: 10.1093/infdis/jit082. Epub 2013 Feb 28. PMID 23448727
- [Derived] Mita-Mendoza NK, van de Hoef DL, Lopera-Mesa TM, Doumbia S, Konate D, Doumbouya M, Gu W, Anderson JM, Santos-Argumedo L, Rodriguez A, Fay MP, Diakite M, Long CA, Fairhurst RM. A potential role for plasma uric acid in the endothelial pathology of Plasmodium falciparum malaria. PLoS One. 2013;8(1):e54481. doi: 10.1371/journal.pone.0054481. Epub 2013 Jan 22. PMID 23349902
- [Derived] Lopera-Mesa TM, Mita-Mendoza NK, van de Hoef DL, Doumbia S, Konate D, Doumbouya M, Gu W, Traore K, Diakite SA, Remaley AT, Anderson JM, Rodriguez A, Fay MP, Long CA, Diakite M, Fairhurst RM. Plasma uric acid levels correlate with inflammation and disease severity in Malian children with Plasmodium falciparum malaria. PLoS One. 2012;7(10):e46424. doi: 10.1371/journal.pone.0046424. Epub 2012 Oct 5. PMID 23071567